CLINICAL TRIAL: NCT01835210
Title: Effect of Acne Vulgaris on Quality of Life of Teenagers Compared to Parent Perceived Effect on Quality of Life
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Jennifer Sorrell, M.D., Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2012-15072; 2012-15072 (Other: IRB)
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Acne; Quality of Life
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Quality of life: Teenager with acne vulgaris This is an observational study, in which the disease of interest is acne vulgaris.

SUMMARY:
Acne vulgaris is a common problem in the adolescent community. Past research has shown that acne affects teenager's self-esteem and mood. However, no research has evaluated the parent perception of their teenager's acne in comparison to the severity of acne and the patient's own reported quality of life. It is hypothesized that parents of teenagers underestimate how much acne vulgaris affects their teenager's skin disease-related quality of life. Also that teenager's perception of the severity of their acne is greater versus their parent's perception. We believe that increased acne severity based on clinician assessment will correlate with worse quality of life. Teenagers between 12 and 17 years old with a diagnosis of acne by a pediatric dermatologist will be enrolled in this study. The study consists of 1 visit, questions regarding demographics, assessment of the teen's acne, the Skindex-Teen quality of life survey (modified for parents), and 2 Likert scales will be completed. In addition, the clinician will score the teen's acne using the standardized Investigator Global Assessment tool. Statistical analysis will compare teen subject answers to the Skindex-Teen with their parent's answers. Also analyzed will be the severity of acne and differences between the clinician IGA score and Skindex-Teen responses

DETAILED DESCRIPTION:
Acne vulgaris is a prevalent problem in the adolescent community, with the literature citing prevalence between 35 to 90% at some stage and some studies showing the prevalence of comedonal acne approaching 100%. Mean age of onset of acne in girls is 11 years and in boys is 12 years. We know that being afflicted with acne places a significant burden on the life of a teenager, and studies have shown diminished quality of life and increased presence of depressive symptoms in teens with acne. Dalgard et al looked at effects of moderate and severe acne on self-esteem and body satisfaction in adolescents. In their study, girls with acne reported significantly higher levels of depressive symptoms, greater feelings of uselessness, and lower self-attitude, sense of pride, self-worth, and body satisfaction compared to girls without acne; a similar tendency was observed in boys. Halvorsen et al performed a cross-sectional questionnaire-based study to evaluate psychological effects of acne in adolescents aged 18-19 years old. They found that in the 14% of participants who had substantial acne- defined as self reported a lot or very much acne, suicidal ideation was twice as frequently reported in girls and three times more frequently reported in boys compared to subjects of either gender with no or a little acne per patient self report. Suicidal ideation was significantly associated with substantial acne with an odds ratio of 1.80. To our knowledge, there has been no research that evaluates parent perception of their teenager's acne in comparison to clinical data points such as investigator global assessment or patient-reported quality of life. Nor have there been data comparing investigator global assessment of acne with patient-reported Likert scale of acne severity. Magin et al looked at 108 patients, of whom 41 had acne and assessed difference in clinician evaluation of acne severity (using the Leeds method as an indicator of severity) compared to patient assessment of acne. They found a moderately poor agreement between objective clinician assessment and patient self-assessment of acne severity (weighted kappa 0.35, with 95% CI 0.1981 - 0.5084). There have been studies as well showing that patients with acne often underestimate the severity of their acne. Smithard A et al studied 317 students aged 14-16 and found that students tended to underestimate their acne severity, with only 66% of patients with mild acne via Leeds scoring self-determining that they had acne. Demircay et al looked at physician's assessment of acne severity, by means of Global Acne Grading System (GAGS) scoring of 0 as none, 1-18 as mild, 19-30 as moderate and > 31 as severe acne. Patient's assessment of acne severity used a 10-point Likert-type scale. Patients were asked how severe their acne was, and 0 denoted "no acne" and 9 denoted "most severe acne that can be imagined". Results of the Likert-type scale were analyzed in four groups: 0 = none, 1-3 = mild, 4-6 = moderate, 7-9 = severe. No correlation was found between physician GAGS scores and any of the patients' own assessments. Smidt et al developed and validated a quality of life index for adolescents with skin disease, using the adult-oriented Skindex and Skindex-16 instruments as models. Skindex-Teen is a 21-item questionnaire, self-administered by the patient and generally is able to be completed in 5 to 10 minutes. The instrument inquires about the patient's perceptions of his/her primary skin condition during the previous 4 weeks. Standardized responses consist of 4-category choices relating to frequency with 0 being never and 4 being all the time. Analysis demonstrated that the refined Skindex-Teen was a valid and effective way of measuring the effects of skin disease in adolescents. A Likert scale is a type of psychometric scale frequently used in psychology questionnaires. On a questionnaire, a Likert scale asks subjects to circle, check or mark the number that most closely correlates to their feelings on a scale.

We speculate that parents of teenagers underestimate how much acne vulgaris affects their teenager's skin disease-related quality of life. By having both the teenage patient and his/her parent independently complete the Skindex-Teen questionnaire at the same time point, we will be able to assess potential differences in how teenagers perceive their acne and how their parents perceive the impact of the teen's acne on quality of life and correlate this with clinical acne severity.

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 17 years of age
* diagnosis of acne by a pediatric dermatologist
* ability to read and understand English
* age appropriate development

Exclusion Criteria:

• developmental delay

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects will be recruited from the pediatric dermatology clinic at Ann and Robert H. Lurie Children's Hospital of Chicago. Teenagers must be between 12 and 17 years old, and have a diagnosis of acne by a pediatric dermatologist.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Teenager's perception of the severity of their acne. | one visit
  Teenagers will complete a Likert scale for assessment of acne severity.

SECONDARY OUTCOMES:
Quality of Life | one visit
  Parents will each complete Skindex-Teen questionnaires to evaluate the teenager's quality of life.
Quality of Life | One visit
  Teenager's will each complete Skindex-Teen questionnaires to evaluate the teenager's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sorrell, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Stathakis V, Kilkenny M, Marks R. Descriptive epidemiology of acne vulgaris in the community. Australas J Dermatol. 1997 Aug;38(3):115-23. doi: 10.1111/j.1440-0960.1997.tb01126.x. PMID 9293656
- [Background] Dreno B, Poli F. Epidemiology of acne. Dermatology. 2003;206(1):7-10. doi: 10.1159/000067817. No abstract available. PMID 12566799
- [Background] Walker N, Lewis-Jones MS. Quality of life and acne in Scottish adolescent schoolchildren: use of the Children's Dermatology Life Quality Index (CDLQI) and the Cardiff Acne Disability Index (CADI). J Eur Acad Dermatol Venereol. 2006 Jan;20(1):45-50. doi: 10.1111/j.1468-3083.2005.01344.x. PMID 16405607
- [Background] Beattie PE, Lewis-Jones MS. A comparative study of impairment of quality of life in children with skin disease and children with other chronic childhood diseases. Br J Dermatol. 2006 Jul;155(1):145-51. doi: 10.1111/j.1365-2133.2006.07185.x. PMID 16792766
- [Background] Dalgard F, Gieler U, Holm JO, Bjertness E, Hauser S. Self-esteem and body satisfaction among late adolescents with acne: results from a population survey. J Am Acad Dermatol. 2008 Nov;59(5):746-51. doi: 10.1016/j.jaad.2008.07.013. PMID 19119094
- [Background] Halvorsen JA, Stern RS, Dalgard F, Thoresen M, Bjertness E, Lien L. Suicidal ideation, mental health problems, and social impairment are increased in adolescents with acne: a population-based study. J Invest Dermatol. 2011 Feb;131(2):363-70. doi: 10.1038/jid.2010.264. Epub 2010 Sep 16. PMID 20844551
- [Background] Magin PJ, Pond CD, Smith WT, Watson AB, Goode SM. Correlation and agreement of self-assessed and objective skin disease severity in a cross-sectional study of patients with acne, psoriasis, and atopic eczema. Int J Dermatol. 2011 Dec;50(12):1486-90. doi: 10.1111/j.1365-4632.2011.04883.x. PMID 22097994
- [Background] Demircay Z, Seckin D, Senol A, Demir F. Patient's perspective: an important issue not to be overlooked in assessing acne severity. Eur J Dermatol. 2008 Mar-Apr;18(2):181-4. doi: 10.1684/ejd.2008.0384. PMID 18424379
- [Background] Smidt AC, Lai JS, Cella D, Patel S, Mancini AJ, Chamlin SL. Development and validation of Skindex-Teen, a quality-of-life instrument for adolescents with skin disease. Arch Dermatol. 2010 Aug;146(8):865-9. doi: 10.1001/archdermatol.2010.161. PMID 20713817